CLINICAL TRIAL: NCT01406834
Title: Treatment for the Mental Health Impact of Killing in War: Augmentation of Existing Evidence-Based Mental Health Interventions
Brief Title: Treatment for the Mental Health Impact of Killing in War
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 11-06004
Record Dates: First submitted 2011-07-19; First posted 2011-08-01 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; Veterans; Killing; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Impact of Killing CBT Treatment — Treatment will include six, one hours sessions with a licensed clinical psychologist or an advanced postdoctoral fellow under the close supervision of a licensed psychologist.

SUMMARY:
The goal of this project is to test the feasibility, acceptability, and efficacy of a treatment module addressing the mental health and functional impact of killing in the war zone.

The investigators will enroll between 12-20 Veterans who have killed in war and have been diagnosed with post-traumatic stress disorder (PTSD) for a pilot study assessing the efficacy of the six-session treatment. Veterans will be randomized either to the treatment or to the waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* Veteran will need to endorse having taken another life in a war zone context
* Have received some prior evidence-based treatment for PTSD

Exclusion Criteria:

* Meet current or lifetime criteria for a psychotic disorder
* Participants in current PTSD treatment will not be excluded;however,if receiving medications they will need to be stabilized on current medications for at least one month.
* If receiving Prolonged Exposure Therapy or Cognitive Behavioral Therapy, individuals will need to wait two weeks after they have completed the treatment to enroll in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Combat veterans
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in psychological symptoms as measured by the Symptom Checklist-90 (SCL-90-R) | Measured at baseline and study completion (week 7)
  A brief multidimensional self-report inventory that screens for nine symptoms of psychopathology and provides three global distress indicators.

SECONDARY OUTCOMES:
Change in killing-related maladaptive cognitions as measured by the Killing Cognitions Scale (KCS) | Measured at baseline and study completion (week 7)
  Assesses killing-related maladaptive cognitions

CONTACTS AND LOCATIONS:
Overall Officials: Shira Maguen, PhD, Principal Investigator — University of California San Francisco/ San Francisco VA Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States